CLINICAL TRIAL: NCT03244592
Title: Development of Minocycline as a Neuroimmune Therapy for Alcohol Use Disorder
Brief Title: Minocycline for Alcohol Use Disorder
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator left institution prior to enrollment of study participants
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K01AA026005 (NIH); K01AA026005 (NIH)
Record Dates: First submitted 2017-07-28; First posted 2017-08-09 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Alcohol Use Disorder; Inflammation; Neurocognitive Dysfunction; Craving; Alcohol Drinking
Keywords: Minocycline
MeSH Terms: conditions — Alcoholism; Inflammation; Cognition Disorders; Alcohol Drinking; cyclopia sequence | interventions — Minocycline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Minocycline (Active Comparator): 200 mg/day
  Interventions: Drug: Minocycline
- Sugar Pill (Placebo Comparator): Matched placebo
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Minocycline — 200 mg/day
  Arms: Minocycline
Drug: Sugar pill — Matched placebo
  Other Names: Placebo
  Arms: Sugar Pill

SUMMARY:
The objective of this proposal is to advance medication development for alcohol use disorder by examining the efficacy and mechanisms of action of minocycline, a neuroimmune modulator, as a potential treatment. This study has important clinical implications, as the available treatments for alcohol use disorder are only modestly effective and testing novel medications is a high research priority.

DETAILED DESCRIPTION:
The research objective of this project is to advance medication development for AUD by conducting a randomized, double blind, placebo-controlled, neuroimaging study to examine the effects of minocycline on neuroinflammation, alcohol cue reactivity, neurocognitive performance, and alcohol use. In the proposed study, non-treatment seeking individuals with a current DSM-5 AUD diagnosis (N = 32) will be randomized to receive either 200 mg of minocycline per day or placebo for 28 days and complete two laboratory sessions. The first laboratory session will be performed immediately before commencing the medication regimen (day 0) and the second will be completed after taking the medication daily for 28 days. Within each laboratory session, participants will complete a cue reactivity paradigm, neurocognitive performance tasks, and a positron emission tomography (PET) imaging session. Neuroinflammation will be assessed by using PET imaging with the radiotracer N-(2,5-dimethoxy-benzyl)-N-(5-fluoro-2-phenoxyphenyl) acetamide, labeled with carbon-11 ([11C]-DAA1106), which binds to the mitochondrial translocator protein, a marker of activated microglia in brain. Additionally, blood samples will be drawn on days 0, 7, 14, 21, and 28 to measure circulating levels of proinflammatory markers and alcohol use over the four weeks of treatment will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 25 - 45
2. Meet DSM-5 diagnostic criteria for an AUD [n.b., only participants with moderate or severe AUD will be enrolled]
3. Drink ≥ 48 standard drinks in a 30-day period before enrollment

Exclusion Criteria:

1. Currently in treatment for AUD, a history of treatment in the 30 days before enrollment, or currently treatment seeking
2. Current (last 12 months) DSM-V diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine
3. Lifetime DSM-V diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
4. Positive urine screen for narcotics, amphetamines, or sedative hypnotics
5. Serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
6. Pregnancy, nursing, or refusal to use reliable method of birth control (if female)
7. A medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes)
8. AST, ALT, or GGT ≥ 3 times upper normal limit
9. Attempted suicide in the past 3 years and/or serious suicidal intention or plan within the past year
10. Currently on prescription medication that contraindicates use of MINO
11. Any other circumstances that, in the opinion of the investigators, compromises participant safety.
12. Claustrophobia
13. Participating in any other research study involving exposure to ionizing radiation in the past year will be excluded if the total cumulative exposure from the past research studies and the current research study would exceed the limits set by the FDA in 21 CFR 361.1. Specifically, the total cumulated dose to the whole body, active blood-forming organs, lens of the eye, and gonads must remain below 5 rems, and the cumulated dose to all other organs must remain below 15 rems. Potential participants who have had exposure to ionizing radiation in the past year will not be allowed to participate if we are unable to obtain proper documentation quantifying the amount of past exposure.
14. Presence of a metal device in the body (e.g., pacemaker, infusion pump, aneurysm clip, metal prosthesis or plate): Those devices could either interfere with the acquisition of the MRI scan of the brain or for whom the MRI scan would pose a potential risk. If participants have a non-removable device in their body, they must acquire and show a document exhibiting the device is MRI-compatible.
15. low affinity rs6971 genotype

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Microglial Activation | Change from baseline after 28 days of medication dosing
  Level of [11C]DAA1106 binding during PET imaging
Cue-Induced Alcohol Craving | Change from baseline after 28 days of medication dosing
  Alcohol Urge Questionnaire (AUQ)
Alcohol consumption | Day 28 of medication dosing period
  Total drinks consumed
Verbal Learning and Memory | Change from baseline after 28 days of medication dosing
  Hopkins Verbal Learning Test
Set-Shifting | Change from baseline after 28 days of medication dosing
  Wisconsin Card Sorting Test
Response Inhibition | Change from baseline after 28 days of medication dosing
  Stop Signal Task
Manipulative Dexterity | Change from baseline after 28 days of medication dosing
  Grooved Pegboard Test
Executive Function | Change from baseline after 28 days of medication dosing
  Digit Symbol Substitution Test
Memory | Change from baseline after 28 days of medication dosing
  Digit Span
Vocabulary | Change from baseline after 28 days of medication dosing
  WAIS Vocabulary
Executive Function | Change from baseline after 28 days of medication dosing
  Rey Complex Figure Copy

SECONDARY OUTCOMES:
Peripheral Proinflammatory Marker levels | At baseline (day zero) and after 7, 14, and 21 and 28 days of medication dosing
  Serum level of cytokines and innate immune receptors
Alcohol Use Disorder Severity | At baseline (day zero) and after 28 days of medication dosing
  Symptom count from the alcohol module for the Structured Clinical Interview for DSM-5

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roche, PhD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No